CLINICAL TRIAL: NCT06177795
Title: I-SCREEN: Increasing Screening for Cancer Using a Randomized Evaluation of EHR-based Nudges
Brief Title: Increasing Screening for Cancer Using EHR-Nudges
Acronym: I-SCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Amol Navathe, Professor of Health Policy and Medicine, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPCC 12022; R33AG068947 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Screening; Mammogram; Behavioral Economics; Prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: For the Penn trial, primary care clinics will be randomized 2:1 to the intervention arm or control arm using covariate-constrained randomization. Patients identified as at high-risk for non-completion of breast cancer screening will be additionally randomized 1:1 at the individual level to receive an additional intensification nudge compared with the multi-component nudge intervention alone. Penn Medicine is expected to enroll approximately 15,000 patients.
  For the UH trial, primary care providers will be randomized 1:1 to the intervention or control arm using covariate-constrained randomization. UH is expected to enroll approximately 6,416 patients.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Penn: Control (No Intervention): Clinics randomized to the control arm will receive standard of care.
- Penn: Intervention (Experimental): Clinics randomized to the intervention arm will receive the toolkit of clinician and patient facing nudges. Patient nudges will be post-visit text message reminders (standard messaging content). Clinician nudges will be default pended orders.
  Interventions: Behavioral: Post-visit patient text messaging; Behavioral: Default pended order
- Penn: High Risk Intensification (Experimental): Patients in the intervention clinics identified as high risk for noncompletion of mammogram will be randomized 1:1 to receive the high risk intensification arm or remain in the standard intervention arm. Patients in the high risk intensification arm will receive an additional bidirectional texting component.
  Interventions: Behavioral: Post-visit patient text messaging; Behavioral: Default pended order; Behavioral: High risk bidirectional post-visit text messaging
- UH: Control (No Intervention): Primary care providers randomized to the control arm will receive standard of care.
- UH: Intervention (Experimental): Primary care providers randomized to the intervention arm will receive default pended orders for a mammogram.
  Interventions: Behavioral: Default pended order

INTERVENTIONS:
Behavioral: Post-visit patient text messaging — Patients will be sent text message reminders 4 days and 14 days after their primary care visit. The message delivered 4-days post-visit will remind the patient that a screening mammogram was recently ordered by their doctor, that appointments have been reserved for them, and to pre-commit to scheduling. The message delivered at 14-days post-visit will remind the patient of their recent screening mammogram order and encourage them to schedule their appointment, if one has not already been scheduled.
  Arms: Penn: High Risk Intensification; Penn: Intervention
Behavioral: Default pended order — A default pended order for a mammogram will be pended to the patient's upcoming primary care encounter and will be visible to the provider during the visit encounter. Clinical staff will have the option of signing the order or dismissing it if they deem it inappropriate for a given patient.
  Arms: Penn: High Risk Intensification; Penn: Intervention; UH: Intervention
Behavioral: High risk bidirectional post-visit text messaging — High risk patients randomized to receive the high risk intensification nudge will receive a bidirectional text messaging component after their visit. This intervention will query the patient about common questions or concerns about breast cancer screening. The bi-directional text messaging intervention will provide additional educational materials based on patient response as well as information about resources to help navigate to screening.
  Arms: Penn: High Risk Intensification

SUMMARY:
In this study, personalized nudges to clinicians and patients will be evaluated to help increase breast cancer screening rates in accordance with USPSTF guidelines among women with a primary care visit, with a particular emphasis on those at high risk for non-completion of cancer screening. In partnership with Penn Medicine (Penn) and Case Western Reserve University-University Hospitals (UH), two complementary, concurrent, 6-month, cluster-randomized, pragmatic trials will be conducted. Those assigned to the intervention arm will receive the following clinician and patient level nudge interventions: clinicians will receive a default pended order for a mammogram in the visit encounter in the EHR (Penn and UH), and patients will receive post-visit text message reminders to encourage them to schedule their mammogram (Penn). Patients identified as high risk for noncompletion will be individually randomized to receive an additional bidirectional text message nudge or the standard text messaging (Penn).

DETAILED DESCRIPTION:
Cancer is a leading cause of mortality in the United States. While strong USPSTF guideline recommendations support appropriate screening for early detection and to avoid preventable deaths, breast cancer screening is often underutilized. Increasing breast cancer screening rates is challenging, in part, because it requires complementary decisions from clinicians (e.g., recommend and counsel patients about screening) and patients (e.g., to internalize risks and choose to complete screening). Presently, the lack of interventions directly targeting both clinicians' and patients' decision-making may underscore the relatively stagnant screening rates in the United States. There is a significant need to develop and scale low-cost interventions that increase breast cancer screening while simultaneously addressing the needs of high-risk patients and reducing disparities. Building upon prior work, the investigators propose to develop and test EHR-based clinician and patient nudges, with an additional intensified nudge to high-risk patients, to help increase screening mammography rates.

This study consists of two complementary and concurrent, cluster-randomized, pragmatic trials to be conducted at Penn and UH.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria to be eligible:

1. Women between 40 and 74 years of age
2. A scheduled new or return (non-urgent/sick) primary care visit at one of the study practices (Penn Trial) or with one of the study primary care providers (UH Trial)
3. Are overdue and eligible for a mammogram per Health Maintenance
4. Does not have a future scheduled mammogram appointment

For the Penn Trial patient intensification nudge, at least one of the following criteria must be met to be considered high risk and randomized to receive the intensification nudge:

1. Medicare Insurance
2. Medicaid Insurance
3. No EHR patient portal account
4. Zero log-ins to EHR patient portal in the previous year

Exclusion Criteria:

Patients will be excluded from the study if:

1. History of bilateral mastectomy
2. Have a mammogram exclusion modifier in Health Maintenance
3. Have no phone number (home or mobile) listed in their chart (Penn Trial only)

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21120 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who complete a screening mammogram within 3 months after the visit | 3 months
  The primary outcome is screening mammogram completion within 3 months after the first eligible primary care visit.

SECONDARY OUTCOMES:
Proportion of patients who complete a screening mammogram within 6 months after the visit | 6 months
  The secondary outcome is screening mammogram completion within 6 months after the first eligible primary care visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Navathe, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Case Western Reserve University/University Hospitals, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania